CLINICAL TRIAL: NCT06032481
Title: Preoperative Scoring System to Predict the Risk of Lymph Node Metastasis in Cervical Cancer
Brief Title: System to Evaluate the Risk of Lymph Node Metastasis Preoperatively in Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Yebin Feng, Director, Fujian Maternity and Child Health Hospital
Other Study IDs: FujianMCHH-Xu01
Record Dates: First submitted 2023-08-26; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery — Patients confirmed cervical cancer were undergone radical hysterectomy with pelvic lymphadenectomy

SUMMARY:
The lymph node status is difficult to be assessed preoperatively, this study aimed to develop a scoring system for predicting the risk of LNM in cervical cancer patients before operation.

DETAILED DESCRIPTION:
Lymph nodes metastasis (LNM) was proved to be a critical risk factor related to the survival to cervical cancer survival. However, preoperative pelvic magnetic resonance imaging (MR) or computed tomography (CT) tests are less sensitive to assess the risk of lymph node metastasis. PET-CT is too expensive and radiative to be widely used in clinical practice. A model was constructed based on clinical indicators to predict lymph node metastasis preoperatively, providing a reference for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cervical cancer
* FIGO stage IB1-IIA1
* Undergone radical hysterectomy with pelvic lymphadenectomy
* Peformed pelvic MRI examination preoperatively

Exclusion Criteria:

* Had distant metastases diagnosed before or during the surgery
* Underwent neoadjuvant radiotherapy preoperatively
* Underwent neoadjuvant chemotherapy preoperatively
* Incomplete or inaccuratemedical records

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 426 patients with cervical cancer who underwent radical resection in China were recruited
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Overall survival | 60 months
  death or loss of follow-up

SECONDARY OUTCOMES:
Risk factors influenced LNM | 60 months
  A multivariable logistic regression analysis was used to analysis the independent factors that contribute to LNM.
The accuracy of the model | 60 months
  The AUC curve was used to assess the discrimination of the scoring system. The comparison between predicted (mean ± SD) and observed rates of LNM was used to test the calibration. The Hosmer-Lemeshow test evaluated the model fit.

CONTACTS AND LOCATIONS:
Overall Officials: Pengming Sun, Ph.D, Principal Investigator — Fujian Maternity and Child Health Hospital

IPD SHARING:
Plan to Share IPD: Undecided